CLINICAL TRIAL: NCT03975829
Title: An Open Label, Multi-center Roll-over Study to Assess Long-term Effect in Pediatric Patients Treated With Tafinlar (Dabrafenib) and/or Mekinist (Trametinib)
Brief Title: Pediatric Long-Term Follow-up and Rollover Study
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDRB436G2401; 2023-509276-42-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2019-05-30; First posted 2019-06-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Diffuse Astrocytoma; Anaplastic Astrocytoma; Astrocytoma; Oligodendroglioma, Childhood; Anaplastic Oligodendroglioma; Glioblastoma; Pilocytic Astrocytoma; Giant Cell Astrocytoma; Pleomorphic Xanthoastrocytoma; Anaplastic Pleomorphic Xanthoastrocytoma; Angiocentric Glioma; Chordoid Glioma of Third Ventricle; Gangliocytoma; Ganglioglioma; Anaplastic Ganglioglioma; Dysplastic Gangliocytoma of Cerebrellum; Desmoplastic Infantile Astrocytoma and Ganglioglioma; Papillary Glioneuronal Tumor; Rosette-forming Glioneuronal Tumor; Central Neurocytoma; Extraventricular Neurocytoma; Cerebellar Liponeurocytoma; Neurofibromatosis Type 1
Keywords: v600-mutation; neuroblastoma; Trametinib; pediatrics; Langerhans Cell Histiocytosis; low grade glioma; plexiform neurofibromas; high grade glioma; dabrafenib; NF-1
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Ganglioneuroma; Ganglioglioma; Neurocytoma; Neurofibromatosis 1; Neuroblastoma; Histiocytosis, Langerhans-Cell; Neurofibroma, Plexiform; Glioma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dabrafenib and/or trametinib (Experimental): Patients in this study may receive one of the following treatments received in the parent study which are:
  * Patients who received monotherapy of either of dabrafenib or trametinib
  * Patients who received combination of dabrafenib and trametinib
    * Patients who discontinued treatment on parent study are still offered to participate in long-term follow-up
  Interventions: Drug: dabrafenib; Drug: trametinib

INTERVENTIONS:
Drug: dabrafenib — dabrafenib oral, twice daily
  Other Names: DRB436
Drug: trametinib — trametinib oral, once daily
  Other Names: TMT212

SUMMARY:
A roll-over study to assess long-term effect in pediatric patients treated with dabrafenib and/or trametinib.

ELIGIBILITY:
Key Inclusion Criteria:

All Subjects:

* Written informed consent, according to local guidelines, signed by the subjects and/or by the parents or legal guardian prior to any study related screening procedures are performed.
* Participation in a Novartis sponsored study such as CTMT212X2101, CDRB436G2201, CDRB436A2102, regardless of current age.
* Parent study (or cohort of parent study) is planned to be closed.
* Subject has demonstrated compliance, as assessed by the investigator, within the parent study protocol requirement(s).
* Willingness and ability to comply with scheduled visits, treatment plans and any other study procedures.

For Subjects Entering the Treatment Period:

* Subject is currently receiving treatment with dabrafenib/trametinib monotherapy or combination within a Novartis Sponsored Drug Development study. Note that subjects who were on the chemotherapy arm of the CDRB436G2201 study are eligible for treatment period of this study only after crossing over into the experimental treatment arm of the CDRB436G2201 study
* In the opinion of the investigator is likely to benefit from continued treatment.

Key Exclusion Criteria:

All Subjects:

- Subject has participated in a combination trial where dabrafenib and/or trametinib was dispensed in combination with another study medication.

For Subjects Entering the Treatment Period:

* Subject has permanently discontinued from study treatment in the parent protocol due to any reason.
* Treatment with dabrafenib and/or trametinib for the subject's indication is approved for marketing and the appropriate dosage form is commercially available and reimbursed in the local country
* Subject currently has unresolved drug related severe toxicities for which dabrafenib and/or trametinib dosing has been interrupted in the parent study. If the subject should meet criteria to resume treatment on the parent protocol then they may be eligible for treatment in this study.

Other protocol-defined inclusion/exclusion may apply.

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2026-11-06 (Estimated); Study Completion 2026-11-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events and Serious Adverse Events (SAEs) | Baseline up to approximately 7 years
  To assess the long-term safety of treatment with dabrafenib, trametinib or the combination.

SECONDARY OUTCOMES:
Percentage of participants with height (measured by cm or in) changes over time | Baseline up to approximately 7 years
  Developmental monitoring: Serial measurements of height will be collected throughout the study
Percentage of participants with weight (measured by kg or lb) changes over time | Baseline up to approximately 7 years
  Developmental monitoring: Serial measurements of weight will be collected throughout the study
Percentage of participants with skeletal maturation (measured by bone age on x-ray or MRI) changes over time | Baseline up to approximately 7 years
  Developmental monitoring: Serial measurements of skeletal maturation will be collected throughout the study
Percentage of participants with sexual maturation (measured by tanner staging criteria) changes over time | Baseline up to approximately 7 years
  Developmental monitoring: Serial measurements of sexual maturation will be collected throughout the study
Percentage of participants with cardiac function (measured by ECG) changes over time | Baseline up to approximately 7 years
  Developmental monitoring: Serial measurements of cardiac function will be collected throughout the study
Clinical Benefit (measured by CT/MRI) | Baseline up to approximately 7 years
  Disease specific clinical benefit, as determined by investigator using institutional standard of care. Investigator will measure tumor response based on the Response Assessment used for the subject in the parent protocol (Response Assessment in Neuro-Oncology (RANO) criteria for solid tumors, RECIST, NF1 Volumetric, Neuroblastoma, or LCH criteria).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (53):
- United States (12):
  - Phoenix Children s Hospital, Phoenix, Arizona
  - Childrens National Hospital, Washington D.C., District of Columbia
  - Nicklaus Childrens Hospital, Miami, Florida
  - Indiana Uni School of Medicine, Indianapolis, Indiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Ctr, New York, New York
  - Cinn Children Hosp Medical Center, Cincinnati, Ohio
  - St Jude Childrens Research Hospital, Memphis, Tennessee
  - Texas Childrens Hospital, Houston, Texas
- Novartis Investigative Site, CABA, Buenos Aires, Argentina
- Australia (2):
  - Novartis Investigative Site, Darlinghurst, New South Wales
  - Novartis Investigative Site, Parkville, Victoria
- Novartis Investigative Site, Brussels, Belgium
- Brazil (2):
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (3):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Czechia (2):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Copenhagen, Denmark
- Novartis Investigative Site, Tampere, Finland
- France (7):
  - Novartis Investigative Site, Rennes, Brittany Region
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
  - Novartis Investigative Site, Villejuif
- Germany (5):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
- Novartis Investigative Site, Petah Tikva, Israel
- Italy (5):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
- Japan (2):
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Osaka
- Novartis Investigative Site, Utrecht, Netherlands
- Novartis Investigative Site, Moscow, Russia
- Spain (2):
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Novartis Investigative Site, Stockholm, Sweden
- United Kingdom (3):
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com